CLINICAL TRIAL: NCT05686057
Title: The Effect of Cardiac Ischemia and Percutaneous Coronary Intervention on the Changes of sST2 Level
Brief Title: sST2 Biomarker Level in Acute/Chronic Coronary Syndrome After Revascularization
Acronym: ST2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Collaborators: South Valley University (Other)
Responsible Party: Principal Investigator, Areej Ahmad Abdullah Tammam Alkhateeb, Lecturer of Cardiology, Assiut University
Other Study IDs: SVU2023
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Myocardial Ischemia; Heart Failure; Coronary Intervention
Keywords: sST2 biomarker; Modified Gensini Score; Revascularization
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure | interventions — Stents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- single vessel diseased patients: sST2 level will be withdrawn at the baseline and after successful PCI
  Interventions: Device: percutanous coronary angiography with stenting
- 2 vessels diseased patients: sST2 level will be withdrawn at the baseline and after successful PCI
  Interventions: Device: percutanous coronary angiography with stenting
- multivessels diseased patients: sST2 level will be withdrawn at the baseline and after successful PCI
  Interventions: Device: percutanous coronary angiography with stenting
- non-ischemic control patients: sST2 level will be withdrawn at the baseline

INTERVENTIONS:
Device: percutanous coronary angiography with stenting — Revascularization will be done by percutanous intervention after assessment of coronary stenosis by diagnostic coronary angiography under local anaesthesia with fluoroscopic guidance in acute/chronic coronary syndrome cases. The severity of stenosis will be done by modified gensini score from angiogram. An sST2 ELIZA test will be done after withdrawal of the cases' samples.
  Groups: 2 vessels diseased patients; multivessels diseased patients; single vessel diseased patients

SUMMARY:
The role of soluble circulating suppression of tumorigenicity 2 biomarker (sST2) in the ischemic heart disease patient is a debatable point. Therefore the aims of this study are to assess the plasma level of sST2 in ischemic heart disease patients versus non-ischemic ones, the acute changes in its level after percutaneous coronary intervention (PCI) and its relation to the severity of ischemia.

DETAILED DESCRIPTION:
A comparison of ischemic patients and non-ischemic controls will be done. The plasma level of sST2 will be withdrawn at baseline and 24-48 hours after the intervention in ischemic group. Then a study ischemic group will be divided into three subgroups; subgroup-1: single vessel disease, subgroup-2: two vessels disease and subgroup-3: multivessels disease. On admission, there will be a significant difference between the group of acute/chronic coronary syndrome cases and controls as regard sST2 plasma level or not. Moreover, the differences between the three ischemic subgroups at the baseline ST2 level will be assessed. The plasma sST2 level after PCI and the correlation between the acute change in pot-PCI sST2 level and the severity of ischemia by Modified Gensini Score (MGS) will be evaluated. The final question that will be answered by this study does the rapid impact of PCI on sST2 level will be mainly related to the severity of ischemia rather than left ventricular function or not.

ELIGIBILITY:
Inclusion Criteria:

* Any patients aged 40 years or more and have the risk factors of ischemic heart disease (IHD) with coronary artery disease symptoms will be included.
* For control subjects should be aged ≥ 40 years old with IHD risk factors including DM and HTN and without any symptoms or signs of cardiac ischemia.

Exclusion Criteria:

* Any patient with heart failure (EF <50%), any patients with rhythm abnormalities including atrial fibrillation, obese patients, structural heart diseases, uncontrolled chronic diseases such as hypertension or diabetes mellitus, any pulmonary artery or parenchymal diseases up to respiratory failure, acute systemic infection or inflammation, and chronic/acute renal diseases.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All middle-old aged patients with IHD risk factors and acute or chronic coronary syndrome manifestations will undergo all routine investigations at baseline and after 24-48 hours of PCI and the levels of sST2 will be assessed for relations to acute changes in left ventricular EF by using 2-dimensional transthoracic echocardiography (2D-TTE) and the degree of ischemia by using Modified Gensini score. At the same time, the level of sST2 in control group with normal all routine diagnostic investigations will be assessed.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
sST2 biomarker level | 24 hours before intervention
  baseline comparison between ischemic heart disease and non-ischemic heart disease-control groups
sST2 biomarker level | 48 hours post percutanous coronary intervention
  follow up of only ischemic heart disease groups of sST2 level changes after intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - South Valley University Hospital, Qina
  - South Valley University, Qina

IPD SHARING:
Plan to Share IPD: No